CLINICAL TRIAL: NCT07044622
Title: Transcutaneous Electrical Nerve Stimulation (TENS) for Intrauterine Device (IUD) Pain
Brief Title: Transcutaneous Electrical Nerve Stimulation (TENS) for Intrauterine Device (IUD) Insertion Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000038467
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Pain
Keywords: IUD; TENS
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TENS (Active Comparator): For the Active TENS group, the device will be set to 80 Hz (hfTENS) and device intensity (0-8) will be titrated to patient comfort, as is the standard protocol for TENS use.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Placebo TENS (Placebo Comparator): For the placebo TENS group, setup will be identical, but the device will not be turned on.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — The TENS 7000 digital TENS unit is a low cost, over the counter, battery operated device with high consumer ratings. The handheld device works by transmitting an electronically generated topical stimulus to a specified area on the body to alter response to pain signals and promote endogenous endorphin release for pain reduction.
  Arms: Active TENS
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — The TENS 7000 digital TENS unit is a low cost, over the counter, battery operated device with high consumer ratings. The handheld device works by transmitting an electronically generated topical stimulus to a specified area on the body to alter response to pain signals and promote endogenous endorphin release for pain reduction.
  Arms: Placebo TENS

SUMMARY:
This study is a double-blind, randomized, placebo-controlled trial to evaluate the use of high frequency TENS for pain control during IUD insertion. Transcutaneous electrical nerve stimulation (TENS) is a relatively low-cost, low-risk, non-pharmacologic intervention for pain management. Previous studies have found that TENS reduces pain associated with other outpatient gynecological procedures. Participants will be randomized in a 1:1 ratio to either active treatment or placebo (placebo TENS) and record pain scores using a 100 mm visual analog scale (VAS) at the time of IUD insertion. The same device will be used for both active and placebo treatment.

DETAILED DESCRIPTION:
The researchers will recruit eligible participants from patients who opt for IUD initiation or replacement during ambulatory care visits at the Center for Women's Health and Midwifery and Yale Family Planning Clinic. Allocation to treatment will be based on a 1:1 blocked randomization scheme. A member of the research/clinical staff other than the provider performing IUD insertion will identify the treatment allocation assigned to the corresponding subject ID. The research staff member will set up the TENS unit accordingly by applying pads to the participant and initiating treatment with the correct settings. When setup is complete, the provider performing the IUD insertion and other clinical staff assisting with the procedure will enter the exam room with no knowledge of TENS treatment assignment to insert the IUD.

REDCap, a HIPAA-compliant, secure web application used for building and managing online surveys and databases, will be used for data collection in this study. Participants will complete three electronic surveys in REDCap during the study. The first survey is a baseline survey to collect demographics as well as medical, obstetric, and gynecologic history and other characteristics prior to the IUD insertion procedure.

IUD insertion will be performed by complex family planning faculty and fellows, as well as OB/GYN residents on their family planning rotation. A research staff member will be within reach of the study participant during the procedure to collect pain scores using a visual analog scale (VAS) presented on an iPad.

The second survey will have a visual analog scale for study participants to rate their pain between 0 and 100 at the following timepoints during IUD insertion:

1. Baseline
2. Immediately after bimanual exam
3. Immediately after speculum insertion
4. If applicable, immediately after IUD removal
5. Immediately after tenaculum placement
6. Immediately after uterine sounding
7. Immediately after IUD insertion
8. 5 minutes after speculum removal

The third survey will ask participants about reflections on their experience with IUD insertion and acceptability of the TENS device, and their past experiences. Clinical Providers who perform the IUD insertion will be asked to take a post IUD insertion survey. This survey will ask questions about the insertion and perceived patient pain.

Participation in the study is expected to only last one day, the day of IUD insertion.

ELIGIBILITY:
Inclusion Criteria Patient Participants:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* English-speaking individual aged 18 years or older.
* Presenting for IUD initiation or replacement during ambulatory care visits to the Yale Family Planning service and Center for Women's Health and Midwifery clinic.
* Opting for either LNG 52mg or copper T380A IUD.

Inclusion Criteria Provider Participants:

* Review of the provider participant study Information Sheet and provision of verbal consent.
* IUD insertion performed by Yale Family Planning and Center for Women's Health and Midwifery clinic faculty and fellows, as well as OB/GYN residents on their family planning rotation, with IUD insertion competency.
* Performing an IUD insertion on a patient participant who meets all patient participant eligibility criteria

Exclusion Criteria Patient Participants:

* Contraindication to IUD initiation
* Current Pelvic Infection
* Distorted Uterine Anatomy (I.e., uterine septum, didelphys, uterine fibroids with cavity length greater than 12mm)
* Pregnancy
* Any other contraindications to IUD insertion as determined by the patient's clinical care staff.
* Exclusionary criteria for study participation
* Current IUD with no visible strings
* Contraindication or allergy to ibuprofen
* History of chronic pain disorder
* Recent opioid use in the previous 30 days
* History of cardiac arrhythmia
* History of heart disease (i.e., atrial fibrillation, congestive heart failure)
* Presence of an implantable device with an electrical discharge (i.e., pacemaker)
* History of epilepsy
* BMI > 50
* History of TENS use
* Planned pain intervention outside standard of care OR pre-procedure use of non-standard pain medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain reported on Visual Analog Scale (VAS) | Day 1 (Day of IUD insertion)
  Pain Visual Analog Scale - full scale from 0-100, higher score indicates higher level of pain.

SECONDARY OUTCOMES:
Post Procedure Surveys | Day 1 (Day of IUD insertion)
  Identify factors other than exposure to TENS associated with higher reported pain, and the acceptability of the TENS device by both patients and providers. Questions answered as yes or no, or on a 4 to 5-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Madden, MD, MPH, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Center for Women's Health and Midwifery, New Haven, Connecticut
  - Yale Family Planning Clinic, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No
Individual participant data meta-analysis for this study will not be done. De-identified individual participant data will be analyzed according to the statistical plan mentioned in the study protocol for manuscript preparation and journal publication. Individual participant data will be shared within the study team. Also, IPD will be shared with the IRB according to institutional guidelines.

REFERENCES:
- [Background] Gero A, Elliott S, Baayd J, Cohen S, Simmons RG, Gawron LM. Factors associated with a negative Patient Acceptable Symptom State (PASS) response with intrauterine device placement: A retrospective survey of HER Salt Lake participants. Contraception. 2024 May;133:110385. doi: 10.1016/j.contraception.2024.110385. Epub 2024 Feb 1. PMID 38307487
- [Background] Hunter TA, Sonalkar S, Schreiber CA, Perriera LK, Sammel MD, Akers AY. Anticipated Pain During Intrauterine Device Insertion. J Pediatr Adolesc Gynecol. 2020 Feb;33(1):27-32. doi: 10.1016/j.jpag.2019.09.007. Epub 2019 Sep 26. PMID 31563628
- [Background] Wu J, Trahair E, Happ M, Swartz J. TikTok, #IUD, and User Experience With Intrauterine Devices Reported on Social Media. Obstet Gynecol. 2023 Jan 1;141(1):215-217. doi: 10.1097/AOG.0000000000005027. Epub 2022 Dec 5. PMID 36473194
- [Background] Svahn S, Niemeyer Hultstrand J, Tyden T, Ekstrand Ragnar M. Contraception use and attitudes: women's concerns regarding hormonal contraception and copper intrauterine devices. Eur J Contracept Reprod Health Care. 2021 Dec;26(6):473-478. doi: 10.1080/13625187.2021.1975267. Epub 2021 Sep 30. PMID 34590968
- [Background] Bracken J, Graham CA. Young women's attitudes towards, and experiences of, long-acting reversible contraceptives. Eur J Contracept Reprod Health Care. 2014 Aug;19(4):276-84. doi: 10.3109/13625187.2014.917623. Epub 2014 Jun 2. PMID 24882426
- [Background] Mody SK, Farala JP, Jimenez B, Nishikawa M, Ngo LL. Paracervical Block for Intrauterine Device Placement Among Nulliparous Women: A Randomized Controlled Trial. Obstet Gynecol. 2018 Sep;132(3):575-582. doi: 10.1097/AOG.0000000000002790. PMID 30095776
- [Background] Lohr PA, Lyus R, Prager S. Use of intrauterine devices in nulliparous women. Contraception. 2017 Jun;95(6):529-537. doi: 10.1016/j.contraception.2016.08.011. Epub 2016 Aug 31. PMID 27591814
- [Background] Pergialiotis V, Vlachos DG, Protopappas A, Vlachos GD. Analgesic options for placement of an intrauterine contraceptive: a meta-analysis. Eur J Contracept Reprod Health Care. 2014 Jun;19(3):149-60. doi: 10.3109/13625187.2014.903238. Epub 2014 May 14. PMID 24828514
- [Background] Shahnazi M, Nikjoo R, Yavarikia P, Mohammad-Alizadeh-Charandabi S. Inhaled lavender effect on anxiety and pain caused from intrauterine device insertion. J Caring Sci. 2012 Nov 28;1(4):255-61. doi: 10.5681/jcs.2012.035. eCollection 2012 Dec. PMID 25276703
- [Background] Nguyen L, Lamarche L, Lennox R, Ramdyal A, Patel T, Black M, Mangin D. Strategies to Mitigate Anxiety and Pain in Intrauterine Device Insertion: A Systematic Review. J Obstet Gynaecol Can. 2020 Sep;42(9):1138-1146.e2. doi: 10.1016/j.jogc.2019.09.014. Epub 2019 Dec 25. PMID 31882291
- [Background] Cimsir MT, Yildiz MS. Could the Valsalva manoeuvre be an alternative to the tenaculum for intrauterine device insertion? Eur J Contracept Reprod Health Care. 2021 Dec;26(6):503-506. doi: 10.1080/13625187.2021.1934442. Epub 2021 Jun 11. PMID 34114522
- [Background] Rahman M, King C, Saikaly R, Sosa M, Sibaja K, Tran B, Tran S, Morello P, Yeon Seo S, Yeon Seo Y, Jacobs RJ. Differing Approaches to Pain Management for Intrauterine Device Insertion and Maintenance: A Scoping Review. Cureus. 2024 Mar 8;16(3):e55785. doi: 10.7759/cureus.55785. eCollection 2024 Mar. PMID 38586685
- [Background] Gemzell-Danielsson K, Jensen JT, Monteiro I, Peers T, Rodriguez M, Di Spiezio Sardo A, Bahamondes L. Interventions for the prevention of pain associated with the placement of intrauterine contraceptives: An updated review. Acta Obstet Gynecol Scand. 2019 Dec;98(12):1500-1513. doi: 10.1111/aogs.13662. Epub 2019 Jun 27. PMID 31112295
- [Background] Lopez LM, Bernholc A, Zeng Y, Allen RH, Bartz D, O'Brien PA, Hubacher D. Interventions for pain with intrauterine device insertion. Cochrane Database Syst Rev. 2015 Jul 29;2015(7):CD007373. doi: 10.1002/14651858.CD007373.pub3. PMID 26222246
- [Background] Babazadeh-Zavieh SS, Bashardoust Tajali S, Haeri SMJ, Shamsi A. Effects of Transcutaneous Electrical Nerve Stimulation on Chronic Pelvic Pain in Women: A Systematic Review and Meta-Analysis. Complement Med Res. 2023;30(2):161-173. doi: 10.1159/000528133. Epub 2022 Nov 21. PMID 36412569
- [Background] Guy M, Foucher C, Juhel C, Rigaudier F, Mayeux G, Levesque A. Transcutaneous electrical neurostimulation relieves primary dysmenorrhea: A randomized, double-blind clinical study versus placebo. Prog Urol. 2022 Jul;32(7):487-497. doi: 10.1016/j.purol.2022.01.005. Epub 2022 Mar 3. PMID 35249825
- [Background] Gonzalez-Mena A, Leiros-Rodriguez R, Hernandez-Lucas P. Treatment of Women With Primary Dysmenorrhea With Manual Therapy and Electrotherapy Techniques: A Systematic Review and Meta-Analysis. Phys Ther. 2024 May 1;104(5):pzae019. doi: 10.1093/ptj/pzae019. PMID 38366860
- [Background] Lerma K, Goldthwaite LM, Blumenthal PD, Shaw KA. Transcutaneous Electrical Nerve Stimulation for Pain Management of Aspiration Abortion up to 83 Days of Gestation: A Randomized Controlled Trial. Obstet Gynecol. 2021 Sep 1;138(3):417-425. doi: 10.1097/AOG.0000000000004502. PMID 34352845
- [Background] Goldman AR, Porsch L, Hintermeister A, Dragoman M. Transcutaneous Electrical Nerve Stimulation to Reduce Pain With Medication Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jan 1;137(1):100-107. doi: 10.1097/AOG.0000000000004208. PMID 33278292
- [Background] Lison JF, Amer-Cuenca JJ, Piquer-Marti S, Benavent-Caballer V, Bivia-Roig G, Marin-Buck A. Transcutaneous Nerve Stimulation for Pain Relief During Office Hysteroscopy: A Randomized Controlled Trial. Obstet Gynecol. 2017 Feb;129(2):363-370. doi: 10.1097/AOG.0000000000001842. PMID 28079781
- [Background] Njogu A, Qin S, Chen Y, Hu L, Luo Y. The effects of transcutaneous electrical nerve stimulation during the first stage of labor: a randomized controlled trial. BMC Pregnancy Childbirth. 2021 Feb 24;21(1):164. doi: 10.1186/s12884-021-03625-8. PMID 33627077
- [Background] Gopalkrishnan P, Sluka KA. Effect of varying frequency, intensity, and pulse duration of transcutaneous electrical nerve stimulation on primary hyperalgesia in inflamed rats. Arch Phys Med Rehabil. 2000 Jul;81(7):984-90. doi: 10.1053/apmr.2000.5576. PMID 10896017
- [Background] Teoli D, Dua A, An J. Transcutaneous Electrical Nerve Stimulation. 2024 Mar 20. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537188/ PMID 30725873
- [Background] Vance CG, Dailey DL, Rakel BA, Sluka KA. Using TENS for pain control: the state of the evidence. Pain Manag. 2014 May;4(3):197-209. doi: 10.2217/pmt.14.13. PMID 24953072
- See also: Long-Acting Reversible Contraception Implants and Intrauterine Devices — https://www.acog.org/clinical/clinical-guidance/practice-bulletin/articles/2017/11/long-acting-reversible-contraception-implants-and-intrauterine-devices
- See also: Patient-Reported Outcomes Measurement Information System Global-10, PROMIS Global-10. APTA — https://www.apta.org/patient-care/evidence-based-practice-resources/test-measures/patient-reported-outcomes-measurement-information-system-global-10-promis-global-10